CLINICAL TRIAL: NCT06507371
Title: Node-sparing Modified Short-Course Radiation Combined With CAPOX and Tislelizumab for MSS Locally Advanced of Middle and Low Rectal Cancer : An Randomized, Prospective, Multicenter, Open-label, Phase III Clinical Trial (mRCAT-III)
Brief Title: Node-sparing Short-Course Radiation Combined With CAPOX and Tislelizumab for MSS Rectal Cancer
Acronym: mRCAT-III
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sir Run Run Shaw Hospital (Other)
Responsible Party: Principal Investigator, Zhangfa Song, Vice president, Sir Run Run Shaw Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SRRS-mRCA-III
Record Dates: First submitted 2024-07-03; First posted 2024-07-18 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Rectal Cancer
Keywords: node-sparing radiation; PD-1; MSS; short-course radioation
MeSH Terms: conditions — Rectal Neoplasms | interventions — spartalizumab; Capecitabine; Oxaliplatin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Treatment Arm (Experimental): Participants will receive 5*5Gy node-sparing modified short-course radiation (radiation targeting the tumor bed without irradiating surrounding tumor-draining lymph nodes) concurrently with CAPOX and tislelizumab regimens: Oxaliplatin, 130mg/m2, intravenous infusion,d1 of each cycle; Capecitabine, 1000mg/m2, PO, BID, d1-14 and tislelizumab, 200mg intravenous infusion d1 of each cycle. CAPOX and tislelizumab repeat every 3 weeks for 4 cycles. After treatment, digital rectal examination, pelvic MRI, endoscopy, and biopsy will be performed to evaluate the tumor regression grade. Patients will receive TME surgery after the chemo-immunotherapy, pCR rate and TRG grade will be evaluated.
  Interventions: Radiation: node-sparing modified short-course radiotherapy; Drug: PD-1 antibody; Drug: Capecitabine; Drug: Oxaliplatin
- Standard Arm (Experimental): Participants will receive 5*5Gy standard short-course radiation (radiation targeting the tumor bed and surrounding tumor-draining lymph nodes) concurrently with CAPOX regimens: Oxaliplatin, 130mg/m2, intravenous infusion,d1 of each cycle; Capecitabine, 1000mg/m2, PO, BID, d1-14. CAPOX repeat every 3 weeks for 4 cycles. After treatment, digital rectal examination, pelvic MRI, endoscopy, and biopsy will be performed to evaluate the tumor regression grade. Patients will receive TME surgery after the chemo-immunotherapy, pCR rate and TRG grade will be evaluated.
  Interventions: Drug: Capecitabine; Drug: Oxaliplatin; Radiation: standard short-course radiotherapy
- Exploration Arm (Other): Participants will receive 5*5Gy standard short-course radiation (radiation targeting the tumor bed and surrounding tumor-draining lymph nodes) concurrently with CAPOX and tislelizumab regimens: Oxaliplatin, 130mg/m2, intravenous infusion,d1 of each cycle; Capecitabine, 1000mg/m2, PO, BID, d1-14 and tislelizumab, 200mg intravenous infusion d1 of each cycle. CAPOX and tislelizumab repeat every 3 weeks for 4 cycles. After treatment, digital rectal examination, pelvic MRI, endoscopy, and biopsy will be performed to evaluate the tumor regression grade. Patients will receive TME surgery after the chemo-immunotherapy, pCR rate and TRG grade will be evaluated.
  Interventions: Drug: PD-1 antibody; Drug: Capecitabine; Drug: Oxaliplatin; Radiation: standard short-course radiotherapy

INTERVENTIONS:
Radiation: node-sparing modified short-course radiotherapy — radiation targeting the tumor bed without irradiating surrounding tumor-draining lymph nodes: 25Gy/5Fx
  Arms: Treatment Arm
Drug: PD-1 antibody — PD-1 antibody (Tislelizumab): 200mg d1 q3w
  Arms: Exploration Arm; Treatment Arm
Drug: Capecitabine — Capecitabine: 1000mg/m2 d1-14 q3w
Drug: Oxaliplatin — Oxaliplatin: 130mg/m2 d1 q3w
Radiation: standard short-course radiotherapy — radiation targeting the tumor bed and surrounding tumor-draining lymph nodes: 25Gy/5Fx
  Arms: Exploration Arm; Standard Arm

SUMMARY:
This is a randomized, prospective, multicenter, open-label, Phase III clinical trial to evaluate node-sparing modified short-course radiation (Radiation targeting the tumor bed without irradiating surrounding tumor-draining lymph nodes) combined with CAPOX and PD-1 Inhibitor (Tislelizumab) compared with standard short-course radiation combined with CAPOX for patients with MSS middle and low rectal cancer. A total of 170 patients will be enrolled in this trial. The primary endpoint is the rate of pathological complete response (pCR). The EFS rate, ORR, organ preservation rate, long-term prognosis, and adverse effects will also be analyzed.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who have a strong willingness to preserve the anus and are willing to receive neoadjuvant therapy.
2. Male or Female aged 18-75.
3. Patients diagnosed with low rectal cancer within 10 cm from the lower edge of the tumor to the anal verge by pelvic MRI and anorectoscopy, the clinical stage is cT3-4bN0/+M0, and the lymph nodes are limited to the mesorectum.
4. Histologically confirmed rectal adenocarcinoma; Genetic testing suggests MSI-L or MSS, or tumor biopsy immunohistochemistry reveals pMMR, that is, MSH1, MSH2, MSH6, and PMS2 are all positive.
5. Eastern Cooperative Oncology Group (ECOG) score 0-1.
6. No previous treatment (including anti-tumor therapy, immunotherapy or pelvic radiation).
7. Laboratory tests indicating no contraindications to radiotherapy, chemotherapy and immunotherapy.
8. Informed consent form signed.

Exclusion Criteria:

1. Patients with a previous history of malignant tumors besides rectal cancer.
2. Patients with distant metastases before enrollment.
3. Patients with positive internal or external iliac lymph nodes are assessed by MRI or CT.
4. Patients with obstruction, perforation, or bleeding that require emergency surgery.
5. Patients with severe concomitant diseases and estimated survival time ≤ 5 years.
6. Allergic to any component of the therapy.
7. Patients who received immunosuppressive or systemic hormone therapy for immunosuppressive purposes within 1 month prior to the initiation of therapy.
8. Patients who have received any other experimental drug (including immunotherapy) or participated in another interventional clinical trial within 30 days before screening.
9. Factors leading to study termination, such as alcoholism, drug abuse, other serious illnesses (including psychiatric disorders) requiring combination therapy, and patients with severe laboratory abnormalities.
10. Patients with congenital or acquired immune deficiency (such as HIV infection).
11. Vulnerable groups, including mentally ill, cognitively impaired, critically ill patients, minors, pregnant or lactating women, illiterate, etc.
12. Other conditions that investigators consider not suitable for this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2024-07-29 (Actual); Primary Completion 2026-02-15 (Estimated); Study Completion 2026-08-15 (Estimated)

PRIMARY OUTCOMES:
pathological complete response (pCR) rate | within 10 days after completion of surgery
  Pathological complete response (pCR) rate

SECONDARY OUTCOMES:
event free survival (EFS) | 3 years after randomization
  the time from randomization until relapse or progression
overall response rate (ORR) | within 10 days after completion of chemotherapy
  The ORR represents the proportion of patients whose tumor burden decreases by a pre-defined clinically meaningful threshold and is maintained for a minimum required duration, which included complete response (CR) rate and partial response (PR) rate
organ preservation rate | within 10 days after completion of chemotherapy
  patients who are able to retain their rectum/anal sphincter after treatment, without requiring a permanent colostomy.
Disease free survival(DFS) | 3 years after chemotherapy or surgery
  The three-year disease-free survival of patients.
Overall survival(OS） | 3 years after chemotherapy or surgery
  The three-year overall survival of patients.
Adverse effects rate | From date of initiation of treatment until the date of death from any cause, assessed up to 5 years
  Rate of radiotherapy, chemotherapy and immunotherapy related adverse events
Rectal specific quality of life assessment via QLQ-CR29 Rectal specific quality of life assessment via QLQ-CR29 Rectal specific quality of life assessment via QLQ-CR29 | Baseline and months 3, 6, 12, 24, 36, 60 after the chemotherapy or surgery
  Rectal specific quality of life according to European Organization for Research and Treatment of Cancer ( EORTC) Quality of life questionnaire QLQ-CR29. scale from 0 to 100, A higher scale represents better function and a higher quality of life.
Quality of life assessment via QLQ-C30 | Baseline and months 3, 6, 12, 24, 36, 60 after the chemotherapy or surgery
  Quality of life according to EORTC Quality of life Questionnaire QLQ-C30 version 3.0. Score range from 0 to 100 points. A higher score represents better function and a higher quality of life
Validation of the Wexner score | Baseline and months 3, 6, 12, 24, 36, 60 after the chemotherapy or surgery
  The change of severity of fecal incontinence assessment according to Wexner score. a score from 0-20, where 0 is perfect continence and 20 is complete incontinence.

CONTACTS AND LOCATIONS:
Locations (1):
- Sir Run Run Shao hospital, Hanzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No